CLINICAL TRIAL: NCT01538264
Title: Blood Flow MRI for Monitoring of Glioma Angiogenesis
Brief Title: Blood Flow MRI for Monitoring Brain Tumors
Acronym: Glioma
Status: Active, not recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Alsop, Professor of Radiology, Beth Israel Deaconess Medical Center
Other Study IDs: 2006P000116; R01CA115745-05 (NIH)
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Brain Tumors
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are studying the use of an advanced magnetic resonance imaging (MRI) technique for measuring blood flow into brain tumors. This technique does not use radioactive tracers, and it can provide high quality images that can be obtained in a standard MRI scanner.

DETAILED DESCRIPTION:
Our goals are:

1. To compare the blood flow measured with this technique with measures of tumor blood vessel density in pieces of the tumor surgically removed as a normal part of clinical treatment. This will confirm a relationship between the imaging measurements and the microscopic characteristics of tumors.
2. To compare the blood flow in tumors before therapy with the concentration of choline, an indicator of cell proliferation. This choline concentration can be measured with another MRI technique. This information will demonstrate the relationship between cell proliferation and blood supply and will also determine whether the choline measurement adds additional information that is clinically necessary.
3. To determine the reproducibility of blood flow measurements in tumors. This is necessary to better understand the sensitivity of the technique to changes in flow caused by a treatment or changes in tumor vascularity.
4. To monitor changes in blood flow after initial treatment. Since sometimes tumors can reappear, the repeated measures will help determine how useful this new imaging technique is at detecting such recurring tumors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with or are suspected of having a glioma

Exclusion Criteria:

* contraindications to MRI which may include the following

  1. Pacemaker
  2. MRI incompatible metal implant
  3. Recently implanted vascular clip
  4. History of claustrophobia
  5. Metal fragment within the eye

Subjects who have received nonstandard therapy may be excluded if the therapy might alter tumor blood flow or other imaging characteristic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects will be brain tumor patients recruited through the Brain Tumor Center at the Beth Israel Deaconess Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2006-06; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David C Alsop, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No